CLINICAL TRIAL: NCT03536728
Title: Phase I Dose-Finding, Safety Study of Oral AMXT 1501 Dicaprate and Difluoromethylornithine (DFMO) in Patients With Advanced Solid Tumors
Brief Title: Oral AMXT 1501 Dicaprate in Combination With DFMO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aminex Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AMXT1501-101A
Record Dates: First submitted 2018-04-04; First posted 2018-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Cancer; Solid Tumor; Solid Carcinoma; Advanced Cancer
Keywords: DFMO; AMXT 1501
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Dose escalation of AMXT1501 with a fixed low dose of DFMO will follow a 3 + 3 dose escalation design. The AMXT 1501 starting dose administered in the first cohort will be 80 mg (2 capsules); each capsule contains 40 mg of active drug. The dose will be given orally, once daily, fasted state alone for 14 days, and starting on Day 15 AMXT 1501 80 mg given in combination with fixed low-dose oral DFMO at 250mg 2x per day (BID), for an additional 14 days; for a total 28 days of treatment per cycle. Cycle 2 includes AMXT1501 + DFMO that will be administered for 28 days. The patient can be treated for additional 28 day treatment cycles as deemed appropriate by their study investigator. Dose escalation of AMXT1501 alone will increase per Part 1 cohort.
  Interventions: Drug: AMXT1501; Drug: DFMO
- Part 2 (Experimental): Dose escalation of DFMO with the Part 1 AMXT1501 RP2D fixed dose will follow a 3 + 3 dose escalation design.
  The AMXT 1501 starting dose administered in the first cohort will be one level below the AMXT 1501 Part 1 RP2D with 500 mg DFMO BID. The morning dose will be given orally of both AMXT1501 and DFMO, in a fasted state. The evening dose of DFMO alone will be given prior to bed-time for 28 days per cycle. The patient can be treated for additional 28 day treatment cycles as deemed appropriate by their study investigator. Dose escalation of DFMO alone will increase per Part 2 cohort.
  Interventions: Drug: AMXT1501; Drug: DFMO
- Expansion (Experimental): The expansion cohort will include up to 14 evaluable patients at a proposed RP2D level of AMXT1501 and DFMO defined by Part 2 to further characterize safety at proposed RP2D dose level with repeat dosing, and characterize early anti-tumor activity.
  Interventions: Drug: AMXT1501; Drug: DFMO

INTERVENTIONS:
Drug: AMXT1501 — AMXT 1501 dicaprate is D-lys(palmitoyl)-spermine dicaprate salt in 40 mg or 200 mg (free base content) enterically-coated capsules
Drug: DFMO — DFMO is DL-2-(difluoromethyl) ornithine monohydrochloride monohydrate 250 mg in hard gelatin capsules
  Other Names: difluoromethyl ornithine monohydrochloride

SUMMARY:
A Phase 1 study will be conducted to establish safety and dose level of AMXT 1501 dicaprate alone, and in combination with DFMO, in cancer patients.

DETAILED DESCRIPTION:
The objective of this study is to determine the safety and tolerability of oral AMXT 1501 dicaprate (AMXT1501) in combination with DFMO in patients with advanced solid tumors. Secondary objectives include characterization of plasma pharmacokinetics (PK) of AMXT 1501 as well as pharmacodynamic (PD) assessment of the impact of AMXT 1501 in combination with DFMO on polyamine uptake by circulating lymphocytes (blood cells).

To these aims, the study will evaluate the safety, PK and PD profiles of orally-administered AMXT 1501 and DFMO. Approximately, 52 patients will be enrolled to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of AMXT 1501 and DFMO in combination. The MTD is defined as the highest dose level below at which dose escalation is stopped.

ELIGIBILITY:
Patient Inclusion Criteria

Individuals eligible to participate in this study must meet all the following criteria:

1. Understand and sign written Institutional Review Board (IRB)-approved informed consent form and be willing to comply with all study procedures.
2. Participants must be ≥18 years of age.
3. Patient is able to take oral medications.
4. Histologically or cytologically documented disease, with the exception of patients with cancers that are not biopsied but where there is radiological evidence of documented disease.
5. Unresectable, locally advanced, or metastatic solid tumor for which no standard therapy is recognized or for which standard therapy has failed.
6. Has evaluable or measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria or mRECIST criteria for pleural mesothelioma (Appendix 2).
7. Tumor tissue and/or archival tissue, ideally from original diagnostic block or the patients most recent biopsy, must be located with plans to be forwarded to the study center or made available prior to the first dose of study therapy and available for biomarker analysis. Archival biopsy samples are only required for patients enrolled in Part 1 or 2.
8. Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale (Appendix 1).
9. Normal auditory acuity: defined as a normal age-related audiogram.
10. Must have adequate bone marrow and renal/hepatic function at the screening and baseline visits, defined as:

    1. Absolute neutrophil count (ANC) ≥1.5×109/L without granulocyte colony stimulating factor (G-CSF) support within 7 days preceding the lab assessment.
    2. Platelet ≥100×109/L, without transfusion within 7 days preceding the lab assessment.
    3. Hemoglobin ≥9 g/dL, without transfusion support within 7 days preceding the lab assessment.
    4. Activated partial thromboplastin time/ partial thromboplastin time (aPTT/PTT) ≤1.5×ULN.
    5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN (if liver metastases are present, then ≤5×ULN is allowed).
    6. Total serum bilirubin ≤1.5×ULN, (except for patients with known Gilbert's Syndrome in whom ≤3×ULN is permitted). Confirmation of Gilbert's diagnosis requires elevated unconjugated (indirect) bilirubin values; normal complete blood count in previous 12 months, blood smear, and reticulocyte count; normal aminotransferases and alkaline phosphatase (ALK) in previous 12 months.
    7. The patient is clinically euthyroid.
    8. Renal: Serum creatinine ≤1.5×ULN or creatinine clearance ≥60 mL/min/1.73m2 for patients with serum creatinine levels above 1.5×ULN.
    9. Any Grade 3 or higher lab abnormalities should be discussed and approved by the Medical Monitor prior to enrollment (even if not considered clinically significant);
11. Patient compliance and geographic proximity (as determined by the PI) that allow adequate follow-up.
12. Both male and female patients must be willing to consent to using highly effective contraception (see Section 9.7.3) prior to study entry, while on treatment and at least 3 months thereafter.
13. Patient with DIPG must:

    a) Be ≥12 years of age and >40 kg in weight. b) Have radiologically documented disease: i. Patient with refractory or progressive DIPG, defined as tumors with a pontine epicenter and diffuse involvement of at least 2/3 of the pons, are eligible without histologic confirmation.

    ii. Patients with brainstem tumors that do not meet radiographic criteria or are not considered to be typical DIPG will be eligible if the tumors have been biopsied and proven to be high-grade gliomas (such as anaplastic astrocytoma, glioblastoma H3K27M mutant DMG).

    c) Have evaluable or measurable disease by magnetic resonance imaging (MRI) criteria (Cooney et al., 2020).

    d) Performance score: i. Patients >16 years of age, Karnofsky score ≥50% (Appendix 5). ii. Patients >12 and ≤16 years of age, Lansky ≥50% (Appendix 6). Note: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

    e) Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy: i. Myelosuppressive chemotherapy: At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea).

    ii. Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor.

    iii. Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.

    iv. Immunotherapy: At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines.

    v. Monoclonal antibodies: >21 days must have elapsed from the infusion of last dose of antibody and toxicity related to antibody therapy must be recovered to Grade ≤1.

    vi. Radiation therapy: Patients must have had their last fraction of craniospinal or focal irradiation >4 weeks prior to enrollment.

    vii. Stem Cell Transplant: Patients must be ≥3 months since autologous stem cell transplant. Patients who received allogenic stem cell transplant or solid organ transplant are not eligible for study.

    Patient Exclusion Criteria

    Individuals will be excluded from study participation if they:

1) Have a seizure disorder where >1 seizure has occurred within the last year. 2) Have clinically significant cardiovascular disease (e.g., significant cardiac conduction abnormalities, uncontrolled hypertension, myocardial infarction, cardiac arrhythmia or unstable angina, New York Heart Association Grade 3 or greater congestive heart failure, serious cardiac arrhythmia requiring medication, Grade 2 or greater peripheral vascular disease, or history of cerebrovascular accident [CVA]) within 6 months of enrollment.

3) History or presence of an abnormal ECG that, in the Investigator's opinion, is clinically meaningful. Screening QTcF interval >480 ms is excluded. In the event that a single QTcF is >480 ms, the patient may enroll if the average QTcF for the 3 ECGs is <480 ms. For patients with an intraventricular conduction delay (QRS interval >120 ms), the JTc interval may be used in place of the QTcF with Sponsor approval. The JTc must be <340 ms if JTc is used in place of the QTcF. Patients with an intraventricular delay due to a left bundle branch block are excluded. Note: QTcF prolongation due to pacemaker may enroll if the JTc is normal.

4) Patient with treated (surgically excised or irradiated) and stable brain metastases are eligible as long as the treatment was at least 4 weeks prior to initiation of study drug and baseline brain computed tomography (CT) with contrast or MRI within 2 weeks of initiation of study drug is negative for new brain metastases. Patients with stable brain metastases must not require therapy with corticosteroids.

5) Have major surgery, other than diagnostic surgery, within 4-weeks prior to Day 1.

6) Have active, bacterial, viral, or fungal infections, requiring systemic therapy.

7) Women who are pregnant or lactating. NOTE: Women of childbearing potential (WOCBP) must have a "negative" serum pregnancy test within 1 week prior to treatment.

a) Women not OCBP defined as any of the following: i. Postmenopausal with >1 year since last menses and:

1. If younger than 65 years old, with a follicle-stimulating hormone (FSH) >40 mIU/mL.
2. If older than 65 years old and not on hormone replacement therapy (HRT), with a FSH >30 mIU/mL.
3. If older than 65 years old and on HRT, the FSH requirement in not applicable. Postmenopausal females on HRT will be allowed if the treatment is stable for at least 6 months prior to dosing of study drug(s).
4. Written medical documentation of being sterilized (e.g. hysterectomy, double oophorectomy, bilateral salpingectomy) with the procedure performed at least 6 months prior to dosing study drug(s). Note: Tubal ligation is not considered a form of permanent sterilization.
5. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

8) Have undergone treatment with radiation therapy, surgery, chemotherapy, or immunotherapy, within 4-weeks prior to study entry (6 weeks for nitrosoureas or Mitomycin C). Patients may also not have any unresolved toxicity >Grade 1 from previous anticancer therapy, except for stable chronic toxicities that are not expected to resolve (i.e. peripheral neuropathy, alopecia etc.). Patients who have an ongoing requirement for thyroid replacement therapy from prior exposure to a checkpoint inhibitor but who are clinically euthyroid are permitted.

9) Have an unwillingness or inability to comply with procedures required in this protocol.

10) Current active liver disease from any cause, including hepatitis A (hepatitis A virus immunoglobulin M positive), hepatitis B (hepatitis B virus [HBV] surface antigen positive), or hepatitis C (hepatitis C virus [HCV] antibody positive, confirmed by HCV ribonucleic acid). Subjects with HCV with undetectable virus after treatment are eligible. Subjects with a prior history of HBV are eligible if quantitative polymerase chain reaction (PCR) for HBV DNA is negative. Note that elevated levels of biotin may interfere with viral serology testing.

11) Have a serious nonmalignant disease that in the opinion of the Investigator and/or the Medical Monitor, could compromise protocol objectives.

12) Patients who are currently receiving any other investigational agent or who have received an investigational agent within the last 28 days.

13) Known gastrointestinal disease or procedure that could interfere with the absorption of study drug, including inability to swallow whole capsules or conditions that may interfere with absorption. The Medical Monitor should be contacted for any questions regarding this exclusion criterion.

14) Patients who have exhibited allergic reactions to a similar structural compound, biological agent, or formulation.

15) Use of biotin (i.e., Vitamin B7) or supplements containing biotin higher than the daily adequate intake of 30 µg (NIH-ODS, 2020). (Note: Subjects who switch from a high dose to a dose of 30 µg/day or less are eligible for study entry.) 16) Infection with human immunodeficiency virus (HIV)-1 or HIV-2. Exception: subjects with well-controlled HIV (e.g., CD4 >350/mm3 and undetectable viral load) are eligible.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Determine DLTs and RP2Ds in AMXT 1501 in combination with DFMO | 2 years
  To evaluate dose-limiting toxicities (DLTs) of AMXT 1501 in combination with DFMO, in patients with advanced cancer and to establish a recommended Phase 2 dose (RP2D)
Determine safety and tolerability of AMXT1501 in combination with DFMO | 2 years
  To evaluate the safety and tolerability of AMXT1501 and DFMO combination

SECONDARY OUTCOMES:
Determine the PK using AUC of AMXT 1501 and in combination with DFMO | 6 months
  To evaluate the pharmacokinetics (PK) of AMXT 1501 alone and in combination with DFMO
Determine the PK using Cmax of AMXT 1501 and in combination with DFMO | 6 months
  To evaluate the pharmacokinetics (PK) of AMXT 1501 alone and in combination with DFMO
Characterize investigator defined response Overall Response Rate (ORR) using RECIST v1.1 | 6 months
  To characterize Investigator defined Overall Response Rate (ORR) using RECIST v1.1 response criteria.
Characterize investigator defined Duration of Response (DOR) | 6 months
  To characterize Investigator defined Duration of Response (DOR), using RECIST v1.1 response criteria and length of time (in days) from last study drug administration to time patient has progressive disease.
Characterize AMXT1501 in combination with DFMO on the expression of immune related gene signatures | 1 year
  Evaluate the effects of treatment with AMXT1501 in combination with DFMO on the expression of immune related gene signatures, immune cell phenotype by IHC, AMXT1501 and DFMO drug levels impact on polyamine levels

OTHER OUTCOMES:
Evaluate AMXT1501 in combination with DFMO on PD biomarker by evaluating the level/concentration of polyamine uptake in the blood. | 6 months
  To evaluate the effect AMXT1501 in combination therapy with DFMO on pharmacodynamic (PD) biomarker of polyamine uptake

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Gallegos, BS, MBA, Study Director — Aminex; Jackie Walling, MBChB PhD, Study Chair — Aminex
Locations (4):
- United States (4):
  - Next Oncology - Austin Midtown, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Next Oncology - San Antonio, San Antonio, Texas
  - Virginia Cancer Center, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piha-Paul SA, Tolcher AW, Vandross AL, Spira AI, Burns MR. Phase I dose-escalation trial of AMXT 1501 dicaprate plus difluoromethylornithine: a dual-agent approach targeting immunosuppressive polyamine metabolism. ESMO Open. 2025 Sep;10(9):105576. doi: 10.1016/j.esmoop.2025.105576. Epub 2025 Sep 6. PMID 40913836